CLINICAL TRIAL: NCT00839956
Title: Bortezomib and Vorinostat as Maintenance Therapy After Autologous Stem Cell Transplant for Multiple Myeloma
Brief Title: Bortezomib and Vorinostat in Treating Patients With Multiple Myeloma Who Have Undergone Autologous Stem Cell Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Leona Holmberg, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2253.00; NCI-2009-01474 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2253; 2253.00 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2009-02-07; First posted 2009-02-10 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-04

CONDITIONS: DS Stage I Plasma Cell Myeloma; DS Stage II Plasma Cell Myeloma; DS Stage III Plasma Cell Myeloma
MeSH Terms: interventions — Bortezomib; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (enzyme inhibitor therapy) (Experimental): Patients receive bortezomib IV on days 2 and 5 and vorinostat PO QD on days 1-14. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bortezomib; Drug: Vorinostat

INTERVENTIONS:
Drug: Bortezomib — Given IV
  Other Names: [(1R)-3-Methyl-1-[[(2S)-1-oxo-3-phenyl-2-[(pyrazinylcarbonyl)amino]propyl]amino]butyl]boronic Acid; LDP 341; MLN341; PS-341; PS341; Velcade
Drug: Vorinostat — Given PO
  Other Names: L-001079038; SAHA; Suberanilohydroxamic Acid; Suberoylanilide Hydroxamic Acid; Zolinza

SUMMARY:
This phase II trial studies the side effects of giving bortezomib together with vorinostat and to see how well it works in treating patients with multiple myeloma who have undergone autologous stem cell transplant. Bortezomib and vorinostat may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving bortezomib together with vorinostat after an autologous stem cell transplant may stop the growth of any cancer cells that remain after transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the toxicity of the use of vorinostat and bortezomib as maintenance therapy after autologous transplant.

SECONDARY OBJECTIVES:

I. Evaluate the median time to disease progression.

II. Evaluate survival.

OUTLINE: Patients receive bortezomib intravenously (IV) on days 2 and 5 and vorinostat orally (PO) once daily (QD) on days 1-14. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Any autologous patient who underwent high dose melphalan (>= 140 mg/m^2) therapy or peripheral blood stem cell (PBSC) rescue for any stage of multiple myeloma and did not participate in another clinical transplant trial whose primary endpoint is also evaluating long-term, disease-free survival, or survival
* Platelet count (transfusion independent) > 75,000 cells/mm^3 and absolute granulocyte count > 1500 cells/mm^3 for 5 calendar days after recovery from high dose therapy
* Consenting for study between 30 days to 120 days after transplant
* Female patient of childbearing potential has a negative serum pregnancy test beta-hCG within 72 hours prior to receiving the first dose of vorinostat
* Female patient is either post-menopausal, free from menses for >= 2 years, surgically sterilized, or willing to use 2 adequate barrier methods of contraception to prevent pregnancy or agrees to abstain from heterosexual activity throughout the treatment on study, starting with visit 1 and for 3 months afterward
* Male patient agrees to use an adequate method of contraception for the duration of the treatment on study and for 3 months afterward

Exclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status >= 2
* A left ventricular ejection fraction less than 45% pre-transplant
* Congestive heart disease with transplant, history of myocardial infarction (MI), history of coronary artery disease, or prolonged corrected QT interval (QTC)
* Total bilirubin greater than 2 mg/ml (unless history of Gilbert's disease)
* Serum glutamic oxaloacetic transaminase (SGOT) or serum glutamic pyruvic transaminase (SGPT) > 2.5 x upper limit of normal (ULN)
* Creatinine clearance < 20 ml/minute, calculated by Cockroft-Gault formula or measured urine
* Cannot give informed consent
* Untreated systemic infection
* Poorly-controlled diabetes mellitus (DM)
* >= grade 3 peripheral neuropathy
* Prior history of human immunodeficiency virus (HIV) positivity with pre-transplant evaluation or known history of hepatitis B or C
* Previous history of hypersensitivity to Bortezomib, boron, or mannitol; known hypersensitivity to the components of study drug or its analogs
* Require therapeutic anticoagulation treatment, especially with coumadin
* Potassium (K) and magnesium (Mg) < normal limits
* Patient who has had chemotherapy, radiotherapy, or biological therapy, within 30 days (42 days for nitrosoureas or mitomycin C) prior to initial dosing with study drug(s) or who has not recovered from adverse events due to agents administered more than 30 days earlier; patients who have received localized consolidation radiation to bone only less than 30 days prior to study entry are allowed
* Patient is currently participating or has participated in a study with an investigational compound or device within 30 days of initial dosing with study drugs
* Patient had prior treatment with an histone deacetylase inhibitor (HDAC) inhibitor (e.g., romidespin [depsipeptide], NSC-630176, MS 275, LAQ-824, belinostat [PXD-101], LBH589, MGCD0103, CRA024781, etc.)
* Patients who have received compounds with HDAC inhibitor-like activity, such as valproic acid, as anti-tumor therapy should not enroll in this study
* Patients who have received such compounds for other indications, e.g. valproic acid for epilepsy, may enroll after a 30-day washout period
* History of central nervous system (CNS) disease
* Symptomatic ascites or pleural effusions
* Patient has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Patient is, at the time of signing informed consent, a regular user (including "recreational use") of any illicit drugs, substance abuse or had a recent history (within the last year) of drug or alcohol abuse
* Patient is pregnant or breast-feeding, or expecting to conceive or father children within the projected duration of the study
* Patient with a history of a prior malignancy with the exception of cervical intraepithelial neoplasia; non-melanoma skin cancer; adequately treated localized prostate carcinoma with prostate-specific antigen (PSA) < 1.0; or who has undergone potentially curative therapy with no evidence of disease for five years, and/or who is deemed at low risk for recurrence by his/her treating physician
* Patient has a history or current evidence of any condition, therapy, or lab abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study or is not in the best interest of the patient to participate
* Patient has a history of a gastrointestinal surgery or other procedures that might, in the opinion of the investigator, interfere with the absorption or swallowing of the study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-02; Primary Completion 2012-08 (Actual); Study Completion 2017-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leona Holmberg, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Bortezomib and Vorinostat): Patients receive bortezomib IV on days 2 and 5 and vorinostat PO QD on days 1-14. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity.
  Bortezomib: Given IV
  Vorinostat: Given PO
Period: Overall Study
Arm/Group | Arm I (Bortezomib and Vorinostat)
Started | 31
Completed | 19
Not Completed | 12
Not completed — Adverse Event | 2
Not completed — Lack of Efficacy | 6
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Arm I (Bortezomib and Vorinostat)
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 9
Age, Continuous [Median (Full Range); unit: years] | 60 [40 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Toxicity as Assessed by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v3.0
Description: The first three months of therapy will be used as the time period in which toxicity will be evaluated and stopping rules for unacceptable toxicity will be implemented. Rules for stopping the study will be based on the rate of withdrawal due to significant toxicity (grade IV, non-hematological, non-metabolic, nonperipheral neuropathy).
Time Frame: The first three months of therapy
Population: No patients met stopping rules for significant toxicity in the first three months of therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Bortezomib and Vorinostat)
Number analyzed (Participants) | 31
Participants | 0

2. Secondary Outcome: Time to Disease Progression in Patients Who Progressed
Description: Patients will be followed for initial response to therapy and for progression of disease. Response criteria will be scored according to International Myeloma Working Group uniform response criteria.
Time Frame: Up to 5 years
Population: One subject withdrew from the study within first week of study therapy and changed to different therapy and is not included in this outcome measure.
Measure: Median (Full Range); unit: years
Arm/Group | Arm I (Bortezomib and Vorinostat)
Number analyzed (Participants) | 30
years | 2.1 [0.33 to 5.3]

3. Secondary Outcome: Survival for All Patients
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Bortezomib and Vorinostat)
Number analyzed (Participants) | 30
Participants | 25

4. Secondary Outcome: Median Follow-up Survival for All Patients
Time Frame: Up to 5 years
Measure: Median (Full Range); unit: years
Arm/Group | Arm I (Bortezomib and Vorinostat)
Number analyzed (Participants) | 30
years | 5.15 [3.4 to 6.5]

ADVERSE EVENTS:
Time Frame: Any adverse event that occurs within 30 days of study treatment
Description: Adverse events grades 3 or higher evaluated.
Arm/Group | Arm I (Bortezomib and Vorinostat)
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 3/31
Other Adverse Events (participants affected / at risk) | 21/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Bortezomib and Vorinostat) (N=31)
Influenza A Infection (Infections and infestations) | 1
Elevated Creatinine Kinase Levels (Investigations) | 1
Anaphylactic reaction (Immune system disorders) | 1 — This event was not study drug related.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Bortezomib and Vorinostat) (N=30)
Neutrophil count decreased (Investigations) | 9
Diarrhea (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 4
Platelet count decreased (Investigations) | 4
Nausea (Gastrointestinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No